CLINICAL TRIAL: NCT06621537
Title: Mental Health Burden and Help-seeking Behavior in the Austrian General Population: from Problem to Psychotherapy in Different Population Groups from a Psychotherapy Science Perspective
Brief Title: Mental Health Burden and Help-seeking Behavior in the Austrian General Population
Status: Completed | Type: Observational
Sponsor: Sigmund Freud PrivatUniversitat (Other)
Collaborators: Danube University Krems (Other)
Responsible Party: Sponsor
Other Study IDs: PTW2024_0926
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Screening
Keywords: general population; Austria; help-seeking behavior; symptom burden
MeSH Terms: conditions — Help-Seeking Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Representative Sample of the Austrian General Population: Sample of the Austriang General Population aged >=14 years representative for age, gender, age x gender, region, education

SUMMARY:
This study investigates the symptom burden and help-seeking behavior in the Austrian general population. Current research shows that mental health in Austria has significantly worsened since the COVID-19 pandemic. Lockdowns, social isolation, and uncertainty about the future have led to increased psychological stress, which has remained elevated even after restrictions were lifted. Vulnerable groups such as young people and individuals with a migration background were particularly affected, often experiencing additional stressors like language barriers, cultural differences, and financial strain. Migrant families frequently face more barriers to accessing mental health services, such as linguistic obstacles, lack of knowledge about the healthcare system, insufficient financial resources, stigmatization of mental illness, and cultural differences in understanding mental health. Research shows that migrants are less likely to seek professional help, instead relying on informal networks or alternative healing methods, leaving many untreated.

Therefore, this study aims to further explore these barriers and the differences in help-seeking behavior between individuals with and without migration backgrounds. A representative sample of the Austrian general population will complete validated questionnaires to assess symptom burden, help-seeking behavior, and self-stigmatization. The study findings will help identify obstacles to accessing psychotherapeutic care and provide insight into improving mental health services, particularly for vulnerable groups.

DETAILED DESCRIPTION:
The research project focuses on the mental health and help-seeking behaviors of the Austrian general population, with a particular interest in vulnerable groups like individuals with migration backgrounds.

The study employs a comprehensive approach by using an online survey targeting a representative sample of the Austrian general population. Key areas of focus include the symptom burden related to psychological disorders and help-seeking behaviors. The survey incorporates a range of standardised validated measurement tools, including: CORE-OM (to assess psychological well-being, symptoms, functionality, and risks), GHSQ (to evaluate help-seeking behavior), SSOSH (to measure self-stigmatization), PHQ-9 (to assess depressive symptoms), GAD-7 (to measure generalized anxiety disorder), ISI-7 (for insomnia severity), PSS-4 (for stress), CAGE (for alcohol misuse), SOEP (for loneliness), and open questions on stressors and resources.

This study will provide insights into the mental health challenges faced by the general population and identify specific barriers to accessing psychotherapeutic care among people with migration backgrounds. These findings will inform future interventions and support mechanisms for these groups. The recruitment process will involve a professional survey agency (Marketagent GmbH), which will ensure a representative sample, including participants aged 14 and above. Participants must have adequate German language skills and reside in Austria. The results will contribute to improving mental health services and addressing disparities in care access.

ELIGIBILITY:
Inclusion Criteria:

* at least 14 years old
* Internet access
* sufficient German skills
* residence in Austria

Exclusion Criteria:

* younger than 14 years old
* no access to the Internet
* lack of German language skills
* residence outside Austria

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: representative sample of the Austrian general population according to age, gender, age x gender, region and education level
Sampling Method: Non-Probability Sample
Enrollment: 2025 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
General Help Seeking Behavior | Once in October 2024
  The General Help-Seeking Questionnaire (GHSQ) is a valdiated standardized tool to assess current intentions to seek help from different sources for different problems. The total score ranges from 10 to 70, with higher scores indicating a greater intention to seek help.
Clincial Outcomes in Routine Evaluation | Once in October 2024
  The Clinical Outcomes in Routine Evaluation - Outcome Measure (CORE-OM) is a common self-report measure of global distress with 34 items all answered on the same five level Likert-type scale asking about the respondents state over the last week. It was originally designed and developed in response to a research funding call from the UK Mental Health Foundation which required that the content must cover domains of well-being (4 items), problems (12 items), functioning (12 items) and risk (6 items). The total score ranges from 0 to 136 (sum of items), with higher scores indicating greater symptom/distress burden. Domain scores range from 0 to 16 (well-being), 0 to 48 (problems and functioning) and 0 to 24 (risk). In addition, means can be calculated by dividing the sum of the items by the number of items in the total score or in the respective domains.

SECONDARY OUTCOMES:
Alcohol Abuse | Once in October 2024
  Symptoms of alcohol abuse will be assessed with a brief screening tool, the so-called CAGE questionnaire.
  The acronym stands for 4 yes/no items constituting the screening test:
  1. Have you ever felt that you ought to Cut down on your drinking?
  2. Have people Annoyed you by criticizing your drinking?
  3. Have you ever felt bad or Guilty about your drinking?
  4. Have you ever had a drink first thing in the morn ing to steady your nerves or to get rid of a hangover (Eye-opener)?
  The total score ranges from 0 to 4, with higher scores indicating a greater degree of problem drinking behaviour.
Insomnia Symptoms | Once in October 2024
  Symptoms of sleeping disorders will be assessed with the brief version of the insomnia severity index (ISI-7). The total score ranges from 0 to 28, with higher scores indicating higher levels of sleep problems.
Depressive Symptoms | Once in October 2024
  Symptoms of depression will be assessed with the 9 item version of the Patient Health Questionnaire (PHQ-9). The total score ranges from 0 to 27, with higher scores indicating greater symptom burden.
Symptoms of Anxiety | Once in October 2024
  Symptoms of anxiety will be assessed with the 7 item version of the general anxiety disorder scale (GAD-7). The total score ranges from 0 to 21, with higher scores indicating greater symptom burden.
Self-stigma | Once in October 2024
  The construct of self-stigma as an important factor in people's decisions not to seek (psycho)therapeutic treatment is assessed using the 10-item Self-Stigma of Seeking Help (SSOSH) scale. The total score ranges from 10 to 50, with higher scores indicating higher levels of self-stigma.
Free text questions on resources and burdens | Once in October 2024
  Two free text questions will elaborate on perceived burdens and resources following a previous study in the Austrian general population.
  1. What is currently bothering you the most?
  2. What helps you most to cope with your problems at the moment?
Perceived Stress Level | Once in October 2024
  The perceived stress level will be assessed with the short version of the perceived stress scale comprising 4 items (PSS-4). The total score ranges from 0 to 16, with higher scores indicating greater symptom burden.
Loneliness | Once in October 2024
  Perceived social isolation is assessed using the three-item loneliness scale (SOEP). The total score ranges from 0 to 12, with higher scores indicating greater social isolation.

CONTACTS AND LOCATIONS:
Locations (1):
- Sigmund Freud Univeristy Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wilson, C. J., Deane, F. P., Ciarrochi, J., and Rickwood, D. (2005). Measuring Help-Seeking Intentions: Properties of the General Help-Seeking Questionnaire. Canadian Journal of Counselling, 39(1), 15-28.
- [Background] Vogel, D. L., Wade, N. G., and Haake, S. (2006). Measuring the self-stigma associated with seeking psychological help. Journal of Counseling Psychology, 53(3), 325-337. https://doi.org/10.1037/0022-0167.53.3.325
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Schaffler Y, Gachter A, Dale R, Jesser A, Probst T, Pieh C. Concerns and Support after One Year of COVID-19 in Austria: A Qualitative Study Using Content Analysis with 1505 Participants. Int J Environ Res Public Health. 2021 Aug 3;18(15):8218. doi: 10.3390/ijerph18158218. PMID 34360512
- [Background] Reinwarth AC, Ernst M, Krakau L, Brahler E, Beutel ME. Screening for loneliness in representative population samples: Validation of a single-item measure. PLoS One. 2023 Mar 16;18(3):e0279701. doi: 10.1371/journal.pone.0279701. eCollection 2023. PMID 36928277
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Kraepelien M, Blom K, Forsell E, Hentati Isacsson N, Bjurner P, Morin CM, Jernelov S, Kaldo V. A very brief self-report scale for measuring insomnia severity using two items from the Insomnia Severity Index - development and validation in a clinical population. Sleep Med. 2021 May;81:365-374. doi: 10.1016/j.sleep.2021.03.003. Epub 2021 Mar 16. PMID 33813233
- [Background] Evans C, Connell J, Barkham M, Margison F, McGrath G, Mellor-Clark J, Audin K. Towards a standardised brief outcome measure: psychometric properties and utility of the CORE-OM. Br J Psychiatry. 2002 Jan;180:51-60. doi: 10.1192/bjp.180.1.51. PMID 11772852
- [Background] Dhalla S, Kopec JA. The CAGE questionnaire for alcohol misuse: a review of reliability and validity studies. Clin Invest Med. 2007;30(1):33-41. doi: 10.25011/cim.v30i1.447. PMID 17716538
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417